CLINICAL TRIAL: NCT01569425
Title: Influence of Meal Timing on Glucose Metabolism and Hyperandrogenism in Lean Women With Polycystic Ovary Syndrome
Brief Title: Meal Timing on Glucose Metabolism and Hyperandrogenism in Lean Women With Polycystic Ovary Syndrome
Acronym: M-PCOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Daniela Jakubowicz, Prof. Daniela Jakubowicz MD, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0048-12-WOMC
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Hyperandrogenism; Insulin Resistance
Keywords: PCOS
MeSH Terms: conditions — Hyperandrogenism; Insulin Resistance | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle counseling (Experimental): Lifestyle counseling, with high calorie breakfast
  Interventions: Other: Dietary intervention
- Life Counseling (Active Comparator): Diet with high calorie dinner
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — High Calorie breakfast and high calorie dinner

SUMMARY:
In obese women with polycystic ovary syndrome (PCOS), weight loss improves insulin resistance and hyperandrogenism, resulting in improvement of clinical symptoms. Weight loss is not required in lean PCOS patients; nevertheless, the influence of meal timing and composition on glucose metabolism and hyperandrogenism may have clinical value. In this study the investigators investigate the effects of two isocaloric diets with different meal timing distribution on insulin resistance and hyperandrogenism in lean PCOS patients.

DETAILED DESCRIPTION:
Insulin resistance and hyperinsulinemia plays a pivotal role in the pathogenesis of polycystic ovary syndrome (PCOS). Hyperinsulinemia stimulates ovarian cytochrome P450c17 alpha activity, in obese and nonobese women with PCOS, thereby increasing serum levels of 17-alpha-hydroxyprogesterone, androgens concentrations, decreasing SHBG and promoting the clinical features of hyperandrogenism.

In women with PCOS, weight loss improves insulin resistance and hyperandrogenism, resulting in improvement of clinical symptoms. Since lean women with PCOS do not have the option of weight loss, it is important to know weather diet composition and meal timing distribution may influence glucose metabolism and hyperandrogenism.

We hypothesized that a timing pattern of increased nutrient intake of protein and carbohydrates in the morning, with decreased caloric intake at night would improve insulin sensitivity and hyperandrogenism in lean women with PCOS.

Objective:The objective of this study is to investigate the effects of two isocaloric diets with different meal timing distribution on insulin resistance and hyperandrogenism in lean PCOS women.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥18 and ≤45 years of age
2. Lean women with PCOS (BMI: ≤ 25 kg/m2)
3. Signed informed consent
4. Exclusion of late-onset adrenal hyperplasia by a fasting serum 17- hydroxy progesterone concentration below 200 ng/dl.
5. Acceptable health based on interview, medical history, physical examination, and laboratory tests (SMA20 and CBC).
6. Not dieting and no change in body weight >10 lb = 4.5 kg within the last 6 months
7. Stable physical activity pattern during the three months immediately preceding study initiation
8. Hyperandrogenemia (elevated free testosterone).
9. Normal liver and kidney function
10. Fasting blood glucose <110 mg/dl.
11. No metabolic disease
12. Usually wakes up between 05:00 and 07:00 and goes to sleep between 22:00 and 24:00.
13. Normal TSH and FT4 levels and serum prolactin
14. Acceptable health based on interview, medical history, physical examination, and laboratory tests

Exclusion Criteria:

1. Diabetes mellitus diagnosed by fasting glucose or a 2-hour OGTT, or fasting glucose > 110 mg/dl
2. Clinically significant pulmonary, cardiac, renal, hepatic, neurologic, psychiatric, infectious, malignant disease (other than skin cancer).
3. Current use of oral contraceptives
4. Serum creatinine level > 1.5 mg/dl
5. Abnormal liver function tests defined as an increase by a factor of at least 2 above the upper normal limit of alanine aminotransferase and/or aspartate
6. Any physiologic or mechanical problems preventing dietary adherence
7. Pregnant or lactating
8. Participating in another dietary program or use of weight-loss medications
9. Documented or suspected history (within one year) of illicit drug abuse or alcoholism.
10. Use of psychotropic or anoretic medication during the month immediately prior to study onset
11. Night or rotating shift work
12. Jet lag during the 2 week period immediately prior to study onset

    -

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-06 (Actual); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
hyperandrogenism | 90 days
  Androgens will be evaluate at baseline and after one of two isocaloric diet that differe in meal timing distribution

SECONDARY OUTCOMES:
glucose metabolism | 90 days
  Glucose metabolism will be evaluated at baseline and after one of two isocaloric diets that differ in meal timing distribution

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Jakubowicz, MD, Principal Investigator — Diabetes Unit E. Wolfson Medical Center Tel Aviv University; Mona Boaz, PhD, Study Director — E. Wolfson Medical Center Tel Aviv University; Julio Wainstein, MD, Study Chair — E. Wolfson Medical Center
Locations (1):
- Daniela Jakubowicz, Holon, Tel Aviv, Israel